CLINICAL TRIAL: NCT02229240
Title: Study GLP111892: Albiglutide Versus Placebo as Add-on to Intensified Basal-Bolus Insulin Therapy in Subjects With Type 2 Diabetes Mellitus
Brief Title: Albiglutide Versus Placebo Added-on to Basal-Bolus Insulin Therapy in Subjects With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was cancelled prior to enrolling any patients
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111892
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Albiglutide; Add-on to basal-bolus insulin therapy; Glucagon-like peptide-1 receptor agonist; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albiglutide (Experimental): Subjects will receive once-weekly subcutaneous injections of albiglutide 30 mg (with forced uptitration to albiglutide 50 mg at Week 4) in addition to intensification of background basal-bolus insulin therapy (with or without metformin) according to predefined titration algorithms.
  Interventions: Drug: Albiglutide
- Matching albiglutide placebo (Placebo Comparator): Subjects will receive once-weekly subcutaneous injections of matching albiglutide placebo in addition to intensification of background basal-bolus insulin therapy (with or without metformin) according to predefined titration algorithms
  Interventions: Drug: Matching albiglutide placebo

INTERVENTIONS:
Drug: Albiglutide — Albiglutide is intended for self-administration as a SC injection. It is provided as a fixed dose of 30 mg of albiglutide or 50 mg of albiglutide in a 0.5 mL injection volume, fully disposable pen injector
  Arms: Albiglutide
Drug: Matching albiglutide placebo — Matching albiglutide placebo will be provided as 0.5-mL injection, fully disposable pen injector system
  Arms: Matching albiglutide placebo

SUMMARY:
This Phase IIIb, randomized, double-blind, parallel-group, placebo-controlled, multicenter, treat-to-target study of 26 weeks treatment duration will evaluate the efficacy and safety of once-weekly albiglutide versus placebo as add-on to intensified basal-bolus insulin therapy (with or without metformin) in subjects with Type 2 Diabetes Mellitus (T2DM). Approximately 450 subjects will be randomly assigned in a 1:1 ratio to 1 of 2 treatment groups: albiglutide + intensified basal-bolus insulin therapy (with or without metformin) or placebo + intensified basal-bolus insulin therapy (with or without metformin. The total duration of a subject's participation will be approximately 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older (inclusive at the time of Screening) with T2DM
* HbA1c >=7.5% and <=10.0% at Screening.
* Currently treated with a basal-bolus insulin regimen (with or without metformin) for at least 3 months before Screening. The subject must be taking the following: Basal insulin (1 or 2 daily injections of neutral protamine Hagedorn insulin, insulin glargine, insulin detemir, or insulin degludec) AND Bolus insulin (at least 2 injections of regular insulin, insulin glulisine, insulin aspart, or insulin lispro); In addition, the total daily dose of insulin must be <=150 units; If taking metformin, a stable dose for at least 8 weeks before Screening. Note: Subject should not have received any other antidiabetic medication within 30 days before Screening (e.g., glucagon-like peptide-1 receptor [GLP-1R] agonist, dipeptidyl peptidase-IV inhibitor, sulfonylurea, or thiazolidinedione). Subjects receiving commercially available premixed basal and prandial insulin are not eligible for this study.
* Body mass index <=40 kilogram (kg) per squaremeter (m^2)
* Thyroid-stimulating hormone (TSH) level is normal or clinically euthyroid as demonstrated by further thyroid tests (e.g., free T4 )
* Female subjects of childbearing potential (i.e., not surgically sterile and/or not postmenopausal) must be practicing adequate contraception (as defined in the protocol) for the duration of participation in the study including the 4-week Posttreatment Follow-up Period.
* Willing and able to comply with all study procedures including intensive insulin administration and performance of frequent SMBG profiles according to the protocol
* Able and willing to provide written informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus
* History of cancer that has not been in full remission for at least 3 years before Screening. (A history of squamous cell or basal cell carcinoma of the skin or treated cervical intra-epithelial neoplasia I or II is allowed)
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Current symptomatic biliary disease or history of acute or chronic pancreatitis
* Severe gastroparesis, i.e., requiring regular therapy within 6 months before Screening
* History of significant GI surgery that in the opinion of the investigator is likely to significantly affect upper GI or pancreatic function (e.g., gastric bypass and banding, antrectomy, Roux en Y bypass, gastric vagotomy, small bowel resection, or surgeries thought to significantly affect upper GI function)
* History of severe hypoglycemia unawareness
* Diabetic complications (e.g., active proliferative retinopathy or severe diabetic neuropathy) or any other clinically significant abnormality (including a psychiatric disorder) that, in the opinion of the investigator, may pose additional risk in administering the investigational product
* Clinically significant cardiovascular and/or cerebrovascular disease within 3 months before Screening including, but not limited to, the following: Stroke or transient ischemic attack; Acute coronary syndrome (myocardial infarction [MI] or unstable angina not responsive to nitroglycerin); Cardiac surgery or percutaneous coronary procedure; Current or history of heart failure (New York Heart Association class III or IV)
* Alanine aminotransferase (ALT) >2.5 × upper limit of normal (ULN) or bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). (Chronic stable hepatitis B and C are acceptable if subject otherwise meets entry criteria and is not on active antiviral treatment [e.g., presence of hepatitis B surface antigen or positive hepatitis C test result within 3 months of Screening])
* Hemoglobin <11 g/dL (<110 gram per liter [g/L]) for male subjects and <10 g/dL (<100 g/L) for female subjects at Screening
* Estimated glomerular filtration rate (eGFR) <=30 mL/minute/1.73 m^2 (calculated using the Modification of Diet in Renal Disease [MDRD] formula) at Screening. Note: As the use of metformin in subjects with varying degrees of renal function may differ from country to country, use of metformin should be in accordance with the metformin product label within the participating country.
* Fasting triglyceride level >750 mg/dL at Screening
* Hemoglobinopathy that may affect proper interpretation of HbA1c
* Known allergy to albiglutide or any product components (including yeast and human albumin), any other GLP-1 analogue, insulin, or other study medication's excipients OR other contraindications (per the prescribing information) for the use of potential study medications (e.g., basal-bolus insulin)
* Use of oral or systemically injected glucocorticoids within the 3 months before randomization or high likelihood of a requirement for prolonged treatment (>1 week) in the 6 months following randomization. However, short courses of oral steroids (single dose or multiple doses for up to 7 days) may be permitted provided these cases are discussed with the medical monitor. Inhaled, intra-articular, epidural, and topical corticosteroids are allowed
* Female subject is pregnant (confirmed by laboratory testing) or lactating
* Receipt of any investigational drug within the 30 days or 5 half-lives, whichever is longer, before Screening, a history of receipt of an investigational antidiabetic drug within the 3 months before randomization, or receipt of albiglutide in previous studies
* Subject that, in the opinion of the investigator, will not benefit from participating in a treat to target study aimed at achieving HbA1c of 7.0%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with severe or documented symptomatic hypoglycemia through Week 26 | Up to Week 26
  Severe hypoglycemia is defined as requiring third-party intervention. Documented symptomatic hypoglycaemia is defined as typical symptoms of hypoglycemia with an accompanying plasma glucose concentration <=70 milligram (mg) per decilitre (dL) (<=3.9 millimole per liter [mmol/L]).
Change from baseline in glycosylated hemoglobin (HbA1c) at Week 26 | Week 26

SECONDARY OUTCOMES:
Change from baseline in body weight at Week 26 and over time | Up to Week 26
Total daily insulin dose, basal insulin dose and bolus insulin dose at Week 26 and over time | Up to Week 26
HbA1c change from baseline in over time | Up to Week 26
Fasting plasma glucose (FPG) change from Baseline at Week 26 and over time | Up to Week 26
Proportion of subjects achieving a HbA1c <7.0% and < 6.5% at Week 26 and over time | Up to Week 26
Percentage of subjects achieving HbA1c <7.0% without weight gain after 26 weeks of treatment | Up to Week 26
Percentage of subjects achieving HbA1c <7.0% without severe or documented symptomatic hypoglycemia after 26 weeks of treatment | Up to Week 26
Percentage of subjects achieving HbA1c <7.0% without weight gain and without severe or documented hypoglycemia after 26 weeks of treatment | Up to Week 26
Number of subjects with non-serious adverse events (AE), serious adverse events (SAE), and AEs and SAEs leading to discontinuation | Up to Week 30
Incidence of hypoglycemic events | Up to Week 30
Assessment of clinical laboratory tests, lipids, vital signs, ECGs and physical examinations | Up to Week 30

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline